CLINICAL TRIAL: NCT03809078
Title: A Pilot Study of 68Ga PSMA 11 PET/MRI and 68Ga RM2 PET/MRI for Biopsy Guidance in Patients With Suspected Prostate Cancer
Brief Title: 68Ga PSMA 11 PET/MRI and 68Ga RM2 PET/MRI for Biopsy Guidance in Patients With Suspected Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-48151; PROS0091 (Other: OnCore); IRB-48151 (Other: Stanford IRB); NCI-2019-00236 (Other: CTRP)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BAY 86-7548; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- 68Ga RM2 first followed by 68Ga PSMA11 (Experimental): Participant will be injected IV with 140 ±20% mBq of 68Ga RM2 and then within two weeks Participant will be injected IV with 3 to 7 mCi of 68Ga PSMA11
  Interventions: Drug: 68Ga RM2; Drug: 68Ga-PSMA-11; Device: Investigational PET scanner coils and software
- 68Ga PSMA11 first followed by 68Ga RM2 (Experimental): Participant will be injected IV with 3 to 7 mCi of 68Ga PSMA11 and then within two weeks Participant will be injected IV with 140 ±20% mBq of 68Ga RM2
  Interventions: Drug: 68Ga RM2; Drug: 68Ga-PSMA-11; Device: Investigational PET scanner coils and software

INTERVENTIONS:
Drug: 68Ga RM2 — PET radiopharmaceutical
  Other Names: 68Ga DOTA Bombesin; BAY86 7548
Drug: 68Ga-PSMA-11 — PET radiopharmaceutical
  Other Names: DFKZ 11; HBED CC PSMA; Heidelberg compound
Device: Investigational PET scanner coils and software — GE Healthcare non-approved PET scanner coils and software

SUMMARY:
The objective of the study is to evaluate 68Ga PSMA 11 PET/MRI and 68Ga RM2 PET/MRI for biopsy guidance in patients with suspected prostate cancer.

DETAILED DESCRIPTION:
Primary Objective: To evaluate 68Ga PSMA 11 PET/MRI and 68Ga RM2 PET/MRI for biopsy guidance in patients with suspected prostate cancer.

Exploratory Objective:

* Correlation of 68Ga PSMA 11 uptake and Gleason score at biopsy
* Correlation of 68Ga RM2 and Gleason score at biopsy

ELIGIBILITY:
Inclusion Criteria:

* Suspected prostate cancer
* Planned prostate biopsy
* Able to provide written consent
* Karnofsky performance status of 50 (or ECOG/WHO equivalent)

Exclusion Criteria:

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam
* Metallic implants (contraindicated for MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duan H, Ghanouni P, Daniel B, Rosenberg J, Thong A, Kunder C, Aparici CM, Davidzon GA, Moradi F, Sonn GA, Iagaru A. A Pilot Study of 68Ga-PSMA11 and 68Ga-RM2 PET/MRI for Biopsy Guidance in Patients with Suspected Prostate Cancer. J Nucl Med. 2023 May;64(5):744-750. doi: 10.2967/jnumed.122.264448. Epub 2022 Nov 17. PMID 36396456

RESULTS

PARTICIPANT FLOW:
Period: First Scan
Arm/Group | 68Ga PSMA11 First Followed by 68Ga RM2 | 68Ga RM2 First Followed by 68Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Scan
Arm/Group | 68Ga PSMA11 First Followed by 68Ga RM2 | 68Ga RM2 First Followed by 68Ga PSMA11
Started | 6 (1 participant withdrew prior to receiving the second scan.) | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 68Ga PSMA11 First Followed by 68Ga RM2 | 68Ga RM2 First Followed by 68Ga PSMA11 | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (4.4) | 55.7 (7.3) | 59.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy Results Correlated With PET Based Imaging Findings
Description: Measure of PET based Biopsy Guidance (ie, prostate uptake on 68Ga PSMA 11 and 68Ga RM2 scans).
Time Frame: Up to approximately 2 hours to complete each scan
Population: Participants who completed both scans and who had biopsy done are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 68Ga PSMA11: 68Ga PSMA11 scan prior to biopsy
- 68Ga RM2: 68Ga RM2 scan prior to biopsy
Arm/Group | 68Ga PSMA11 | 68Ga RM2
Number analyzed (Participants) | 13 | 13
Participants | 13 | 13

ADVERSE EVENTS:
Time Frame: 2 weeks, plus safety follow up at to 72 hours after the final scan
Description: One participant discontinued the study prior to receiving the scan using 68Ga RM2.
Arm/Group | 68Ga PSMA11 | 68Ga RM2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03809078/Prot_001.pdf